CLINICAL TRIAL: NCT04978571
Title: A Prospective Study on the Effect of Auricular Percutaneous Electrical Nerve Field Stimulation (PENFS) in Patients With Post Concussion Syndrome (PCS)
Brief Title: Percutaneous Electrical Nerve Field Stimulation (PENFS) in Patients With Post Concussion Syndrome (PCS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Orange County (Other)
Collaborators: Innovative Health Solutions (Industry)
Responsible Party: Principal Investigator, Ashish Chogle, Principal Investigator, Children's Hospital of Orange County
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 190667
Record Dates: First submitted 2021-04-21; First posted 2021-07-27 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Post-Concussion Syndrome; COVID Long-Haul; COVID-19
MeSH Terms: conditions — Post-Concussion Syndrome; Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: Concussion: prospective, randomized-controlled treatment trial. COVID: prospective, open label, non-randomized-controlled treatment trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Concussion: After study completion, a designated member of the study will disclose study group. This designated member will not have direct contact with study participants during their participation.
  COVID: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Active Neurostim Device (Experimental): Patients in this group will receive the active devices for the initial 4 study weeks.
  Interventions: Device: percutaneous electrical nerve-field stimulation, PENFS
- Sham Neurostim Device (Sham Comparator): Patients in this group will receive the sham devices for the initial 4 study weeks. However, they will be offered the 4 active devices after.
  Interventions: Device: percutaneous electrical nerve-field stimulation, PENFS (sham device)
- COVID Active Neurostim Device (Experimental): Patients in this group will receive the active devices for the 6 study weeks.
  Interventions: Device: percutaneous electrical nerve-field stimulation, PENFS (COVID active device)

INTERVENTIONS:
Device: percutaneous electrical nerve-field stimulation, PENFS — A novel, FDA approved for commercial use, cleared device that delivers field stimulation with alternating frequencies to the external ear
  Arms: Active Neurostim Device
Device: percutaneous electrical nerve-field stimulation, PENFS (sham device) — A novel, FDA approved for commercial use, cleared device that delivers field stimulation with alternating frequencies to the external ear. The sham device will not deliver field stimulation to the ear.
  Arms: Sham Neurostim Device
Device: percutaneous electrical nerve-field stimulation, PENFS (COVID active device) — A novel, FDA approved for commercial use, cleared device that delivers field stimulation with alternating frequencies to the external ear
  Arms: COVID Active Neurostim Device

SUMMARY:
The purpose of this study is to test the effect of Auricular Percutaneous Electrical Nerve Field Stimulation (a Neurostim device) on children with pain and Post Concussion symptoms.

An additional purpose of this study is to demonstrate that PENFS improves functioning in children with post Covid-19 symptoms.

DETAILED DESCRIPTION:
The purpose of this study is to test the effect of Auricular Percutaneous Electrical Nerve Field Stimulation (a Neurostim device) on children with pain and Post Concussion symptoms. Patient will be offered a Neurostim device. This device is placed on the outer ear through tiny needles. Since this is a randomized trial, patients may receive an active (experiment) or nonactive (control) Neurostim device. However, the nonactive control Neurostim device group will be given the option to receive an active device after the initial study procedures. The experiment group may be in this study up to 8 weeks and the control group may be in this study up to 12 weeks. The control group will have 4 additional weeks due to the transition to an active device following the first 8 weeks. The device is worn weekly for 4 weeks. Each device is worn for 5 consecutive days for the full 24 hours. The participant will be able to easily take the device off on the 6th day. Study procedures include: Neurological testing- a balance test and computerized neurological standard testing, Cardiology testing- electrocardiogram for heart rate variability (heart electrical pulse test), a pupilometer (eye) test, and parent/child questionnaires. You may benefit from this research, but there is no guarantee that being in this study will help you.

Patients in the COVID arm will be offered 6 placements of Neurostim devices. This device is placed on the outer ear through tiny needles. Patients in this arm will not be randomized, all patients will receive active devices. This group will be in the study for up to 10 weeks. The device is worn weekly for 6 weeks. Each device is worn for 5 consecutive days for the full 24 hours. The patient will be able to remove the device on the 6th day. Study procedures include: Neurological testing called Cognigram to measure cognitive functioning and parent/child questionnaires. After 6 weeks of device placements, parent and child will complete a 1-week and 1-questionnaires. You may benefit from this research, but there is no guarantee that being in this study will help you.

ELIGIBILITY:
Concussion:

Inclusion Criteria:

* Clinical diagnosis of Post-Concussion Syndrome
* Post-Concussion Symptoms for at least 3 months along with lack of other explanation for their symptoms
* English and Spanish-speaking families

Exclusion Criteria:

* Seizure disorders
* Significant developmental delay
* Infection or severe dermatological condition of ear
* Bleeding disorders
* Implanted electrical device

COVID:

Inclusion Criteria

* Child is in between the ages 11-18
* Child is present at CHOC Neurology clinic post covid-19 symptoms of more than 3 months duration along with lack of other explanation for their symptoms
* English-speaking and Spanish-speaking families

You cannot participate in this study if you meet the following exclusion criteria:

* Children with significant developmental delay, infection or severe dermatological condition of ear, bleeding disorders, or having any implanted electrical device will be excluded.
* Are not able to attend Friday appointments for the Neurostim placements.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Immediate Post-Concussion Assessment | 8 weeks
  With the Immediate Post-Concussion Assessment, percentiles indicate functioning assessment after a concussion. Having a higher score on this assessment implies having a worse outcome assessment.
Post-Concussion Symptom Scale | 8 weeks
  Post Concussion Symptom Scale- a 22 item questionnaire, rated on a 0-6 scale. Having a higher score indicates having worse symptom assessment.
Balance Error Scoring Symptom | 8 weeks
  Balance Error Scoring Symptom- a balance test conducted in person. Patient is asked to do a 3 poses on the floor and 3 poses standing on a foam and asked to stand still. The amount of errors will be counted for the times the patient moves. The higher the errors, means patient does not have a well-balance.
COGNIGRAM | 10 weeks
  COGNIGRAM is a test prescribed by clinicians to measure cognitive function.

SECONDARY OUTCOMES:
Abdominal Pain Index | 8 weeks
  4 item to rate abdominal pain. Higher score indicates having worse outcome.
Baxter Animated Retching Faces Nausea Scale | 8 weeks
  rate on a 1-10 scale level of nausea. Higher score indicated feeling worse.
Children's Somatization inventory | 8 weeks
  23 item to rate symptoms, higher score indicates worse symptoms
Functioning disability inventory | 8 weeks
  15 item, asking on functioning, higher score indicated worse outcome.
Patient-Reported Outcomes Measurement Information System- Anxiety | 8 weeks
  8 item questionnaire asking on anxiety level. Higher score indicates worse outcome.
Patient-Reported Outcomes Measurement Information System- Depression | 8 weeks
  8 item asking on depression, higher score indicated worse outcome
Patient-Reported Outcomes Measurement Information System-Global health scales | 8 weeks
  7-item asking on general health, lower score indicates worse outcome
Covid-19 questionnaire | 10 weeks
  40-item asking Covid related symptoms and history.

OTHER OUTCOMES:
Orthostatic Vitals | 8 weeks
  numerical number that determines blood pressure. Having a high blood pressure indicates worse outcome. Reading will be done by a provider.
Electrocardiography | 8 weeks
  Heart rate measurement- a recording of electrical signal from the heart to check for heart conditions. Reading will be done by a provider.
Pupillometry | 8 weeks
  Pupillometry: An eye assessment to measure pupil size and reactivity, reading will be done by a provider

CONTACTS AND LOCATIONS:
Locations (1):
- CHOC Children's, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No